CLINICAL TRIAL: NCT02501057
Title: HealthCall: Enhancing Brief Intervention for HIV Primary Care Alcohol Dependence
Brief Title: Reducing Alcohol Dependence Among HIV-Positive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Deborah Hasin, Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AA023163-01 (NIH)
Record Dates: First submitted 2015-07-13; First posted 2015-07-17 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Dependence
Keywords: Human Immunodeficiency Virus; Unsafe Drinking; Antiretroviral Therapy (ART)
MeSH Terms: conditions — Alcoholism; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clinician's Guide (Active Comparator): The Baseline intervention includes a brief meeting (20 minutes or less) with a clinic staff member to discuss drinking and HIV medication adherence. The clinic staff member provides feedback on the participant's drinking, helps the participant set a drinking goal, and make suggestions to help the participant reduce their drinking. Participant receives a booklet called "Rethinking Drinking" that includes information about alcohol and tips for cutting down on alcohol use or quitting drinking. 30- and 60-day visits last about 10 minutes each, and include a meeting with the clinic staff member again to discuss drinking and HIV medication adherence, and to get additional feedback.
  Interventions: Behavioral: Clinician's Guide
- Enhanced Motivational Interviewing (Active Comparator): Participants meet with a counselor to discuss their alcohol use, the impact it has on their health, and the possibility of reducing their drinking. The first counseling session is intended to help participants reduce their alcohol use. They are asked to describe the pros and cons of their alcohol use and whether it might be important to reduce or quit drinking. After, they are given a study smartphone and asked to use HealthCall-S daily to help keep track of their drinking. At 30 days, participants review a graph showing the results of HealthCall-S use and discuss it with the counselor. They also have a brief discussion about drinking patterns and goals for reduction. They are then asked to continue using HealthCall-S for the next 30 days, after which the counselor meets with the participant for another brief interview to go over the updated graph, and to discuss their experience with HealthCall-S. They will also have a brief discussion about drinking patterns and goals for reduction.
  Interventions: Behavioral: Enhanced Motivational Interviewing
- Enhanced Clinician's Guide (Experimental): Participants in this group receive the Clinician's Guide intervention paired with daily use of HealthCall-S, which includes two cycles of daily use of HealthCall for 30 days, followed by personalized feedback in the form of a graph with a clinic staff member.
  Interventions: Behavioral: Enhanced Clinician's Guide

INTERVENTIONS:
Behavioral: Clinician's Guide — An evidence-based, NIAAA-advocated approach to brief intervention for heavy drinking in primary care settings.
  Arms: Clinician's Guide
Behavioral: Enhanced Motivational Interviewing — Brief motivational interview plus the use of a smart phone application to monitor alcohol use and health behaviors.
  Arms: Enhanced Motivational Interviewing
Behavioral: Enhanced Clinician's Guide — An evidence-based, NIAAA-advocated approach to brief intervention for heavy drinking in primary care settings plus the use of a smart phone application to monitor alcohol use and health behaviors.
  Arms: Enhanced Clinician's Guide

SUMMARY:
The purpose of this study is to compare the effects of interventions for drinking-reduction and antiretroviral therapy (ART) adherence among HIV-positive primary care patients. The interventions consist of brief meetings to discuss drinking and ART adherence enhanced with daily self-monitoring through the use of a smart phone application that tracks drinking and other aspects of health. These meetings will either be based on the Clinician's Guide, a brief intervention for heavy drinking in primary care settings advocated by the National Institute on Alcohol Abuse and Alcoholism, or Motivational Interviewing. Participants will be assessed at baseline, 30, 60, 90 days, 6 and 12 months after baseline. By the end of treatment (60 days) and throughout the follow-up period, alcohol use is expected to highest among participants who receive the Clinician's Guide alone, intermediate among participants who receive the enhanced Clinician's Guide, and lowest among participants who receive enhanced Motivational Interviewing.

DETAILED DESCRIPTION:
HIV infection is a widespread health problem in the U.S. Antiretroviral (ART) therapy has increased longevity and changed the nature of risk factors for morbidity and mortality. Alcohol consumption has become an increasingly serious health issue among HIV primary care patients. Drinking is a key factor in progression to severe liver damage (especially those co-infected with hepatitis), and liver disease is now one of the most common causes of death among those with HIV. Excess drinking is also associated with medication noncompliance, reduces the effect of antiretroviral treatment, and is linked to other health problems. Therefore, helping HIV patients reduce unsafe drinking is crucial to their long-term health. This study aims to evaluate two evidence-based approaches when combined with an innovative smart phone application designed to help users track drinking and other aspects of health. An effective, easily implemented alcohol-reduction intervention could be incorporated into standard care in HIV clinics to help prevent or slow the progress of some medical problems in HIV-infected individuals, improve medication compliance, prolong lifespan and decrease risk behavior associated with alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patient had 4 or more drinks on any day in prior 30 days
* Patient meets criteria for DSM-IV current alcohol dependence
* HIV+

Exclusion Criteria:

* Patient is psychotic, suicidal, or homicidal
* Patient has gross cognitive impairment
* Patient does not speak English or Spanish
* Patient has plans to leave the greater New York metropolitan area within the study period
* Patient has vision/hearing impairment that would preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption in the last 30 days, assessed at baseline and repeatedly during follow-up so that change can be analyzed. | Baseline, 30, 60 days (end-of-treatment), 3, 6, 12 months
  As measured by number of drinks per drinking day and percentage of days abstinent.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah S Hasin, Ph.D., Principal Investigator — Columbia University